CLINICAL TRIAL: NCT02341833
Title: Effects of Preconditioning With Sevoflurane During Organ Procurement From Brain Dead Donors: Impact on Early Function of Liver Allografts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gregory Minguet, Doctor, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-26-06
Record Dates: First submitted 2014-06-26; First posted 2015-01-19 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Post-transplantation Liver Allograft Function
Keywords: Anesthetic preconditioning; Sevoflurane; Liver transplantation; brain-death donors
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Sevoflurane (Active Comparator): 1 MAC of sevoflurane for 15 minutes before organs procurement.
  Interventions: Drug: Sevoflurane
- No intervention (No Intervention): No volatile anesthetics during organs procurement

INTERVENTIONS:
Drug: Sevoflurane — In the sevoflurane group, the anesthetic agent has to be administered immediately after arrival in the operating room to reach an end-expiratory target concentration of 2%. This concentration of sevoflurane should be maintained until the procedural cardiac arrest and for at least 15 min.
  Arms: Sevoflurane

SUMMARY:
The aim of the investigators study is to investigate the effects of anaesthetic preconditioning with sevoflurane during organs harvesting in brain dead donors. More particularly, the investigators will investigate whether sevoflurane preconditioning protects against ischaemia-reperfusion the livers and kidneys allografts after a prolonged period of cold ischaemia and whether this protection translates in a better clinical functional recovery of these allografts.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive brain dead donors in the Belgian university hospitals of Leuven, Brussels, Louvain and Liège eligible for organs harvesting followed by organs transplantation in the Eurotransplant area. There is no age limitation for eligibility

Exclusion Criteria:

* haemodynamic instability that precludes safe administration of 2% sevoflurane.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of liver function following liver transplantation. | First week post-transplantation
  * Transaminases, bilirubin, prothrombin time (PT) and international normalized ratio (INR) on the first post-transplantation blood test and on the following samples from the 1st to the 7th postoperative days.
  * Number of liver recipients that will meet the criteria for "early allograft dysfunction" as defined by :
    * bilirubin ≥10 mg/dL on the 7th day.
    * INR ≥ 1.6 on the 7th day.
    * ALAT or ASAT > 2000 UI/L during the first 7 postoperative days.

SECONDARY OUTCOMES:
• Incidence of primary non function (liver failure requiring emergent re-transplantation) | 30-day and 6-month after transplantation.
• Hospital length of stay. | 30-day and 6-month after transplantation.
• Allograft function (yes/no) at 30-day and 6-month after transplantation. | 30-day and 6-month after transplantation.
• Hospital mortality and at 30-day. | 30-day.

OTHER OUTCOMES:
Composite outcome of post transplantation kidney function. | First week after transplantation, 30 day and 6-month.
  • Creatinine on the first post-transplantation blood test and on the following samples from the first to the 7th postoperative days. Maximal creatinine values and values at 72-hour after transplantation, the time for 50% decline, and the area under the curve during the first postoperative week.
• Delayed graft function : (defined as dialysis during first postop wk; decline in creatinine value | First week after transplantation, 30 day and 6-month.
  * Dialysis during the first postoperative week.
  * Decline in creatinine value of less than 10% per day during 3 consecutive days.
• Length of delayed graft function. | First week after transplantation, 30 day and 6-month.
• Primary non function (patient who must go back to chronic hemodialysis and must be listed for re-transplantation | First week after transplantation, 30 day and 6-month.
  patient who must go back to chronic hemodialysis and must be listed for re-transplantation, at 30-day and 6-month after transplantation.
• Hospital length of stay. | First week after transplantation, 30 day and 6-month.
• Hospital mortality and mortality at 30-day. | First week after transplantation, 30 day and 6-month.

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Joris, MD, PhD, Principal Investigator — CHU Liège - Belgium
Locations (1):
- Department of Anesthesiology, CHU Liège, Liège, Belgium